CLINICAL TRIAL: NCT03877146
Title: Calming Alternatives Learned During MRI-Guided Breast Biopsy (CALM)
Brief Title: Calming Alternatives Learned During MRI-Guided Breast Biopsy
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100029
Record Dates: First submitted 2019-02-26; First posted 2019-03-15 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer; Breast Pain; Pain, Acute; Anxiety; Coping Skills; Self Efficacy
Keywords: Controlled Breathing; MRI-Guided Breast Biopsy; Breast Pain; Body Pain; Anticipatory Pain; Anxiety; Coping Skills; Self Efficacy
MeSH Terms: conditions — Breast Neoplasms; Mastodynia; Acute Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Both conditions receive audio-recordings, and the radiologist care providers are blinded to the audio recordings participants receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control Condition (No Intervention): As part of usual care, participants will be provided with headphones to listen to music during the biopsy procedure. Music options will include instrumental jazz, classical piano, harp and flute, and world music.
- Controlled Breathing Intervention (Experimental): Participants in the controlled breathing intervention will be provided with headphones to listen to the guided intervention audio file. Over the course of the 25-60-minute procedure, approximately 50% of the intervention will be spent completing controlled breathing. The other 50% of the intervention will be spent listening to music, which is part of usual care. Music options will include instrumental jazz, classical piano, harp and flute, nature sounds, and world music.
  Interventions: Behavioral: Controlled Breathing Intervention

INTERVENTIONS:
Behavioral: Controlled Breathing Intervention — Participants in the controlled breathing intervention will be provided with headphones to listen to the guided intervention audio file. The intervention will guide participants to breathe at a rate of six breaths per minute (approximately 50% of their normal breathing rate).
  Arms: Controlled Breathing Intervention

SUMMARY:
The proposed randomized study evaluates whether a controlled breathing intervention could be efficacious for reducing pain in the MRI-guided breast biopsy setting. Support for this intervention stems from experimental and clinical studies on the effects of controlled breathing on pain. Implementing a controlled breathing intervention during MRI-guided breast biopsy has the potential to provide effective pain management in this outpatient setting. The primary study objectives are to assess the feasibility, acceptability, and efficacy of a novel audio-recorded controlled breathing intervention for reducing breast and body pain in women undergoing MRI-guided breast biopsy. The secondary study objectives are to evaluate the effects of controlled breathing on measures of physiological reactivity (i.e., blood pressure and heart rate), pain catastrophizing, and self-efficacy for pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing MRI-guided core needle breast biopsy at the Duke Cancer Institute
* Ability to speak and read in English
* Age ≥ 18 years
* Ability to provide meaningful consent

Exclusion Criteria:

* Hearing impairment that is documented in the medical record that would limit the use of the guided intervention or music
* Cognitive impairment that is documented in the medical record or results in being unable to provide meaningful consent
* Undergoing IV-administered sedation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be women undergoing MRI-guided breast biopsies at the Duke Cancer Institute.
Enrollment: 58 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Body pain pre-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | Baseline
  Body pain pre-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average body pain during the past week, as well as 4) current body pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.
Breast pain pre-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | Baseline
  Breast pain pre-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average breast pain during the past week, as well as 4) current breast pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.
Body pain after positioning on the MRI table: Numerical rating scale (NRS) | After positioning on the MRI table, within 1 minute
  Body pain after positioning on the MRI table for the biopsy procedure will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Breast pain after local anesthetic injection: Numerical rating scale (NRS) | After each superficial local anesthetic injection, within 1 minute
  Breast pain after each superficial local anesthetic injection during the biopsy procedure will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Breast pain after deeper local anesthetic injection: Numerical rating scale (NRS) | After each deeper local anesthetic injection, within 1 minute
  Breast pain after each deeper local anesthetic injection during the biopsy procedure will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Body pain after introducer insertion: Numerical rating scale (NRS) | After last introducer insertion, within 1 minute
  Body pain after the last introducer is inserted will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Breast pain after tissue sampling: Numerical rating scale (NRS) | After last tissue sampling at each biopsy site, within 1 minute
  Breast pain after the last tissue sampling at each biopsy site will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Body pain after introducer sheath removal: Numerical rating scale (NRS) | After last introducer sheath removal, within 1 minute
  Body pain after the last introducer sheath is removed will be will be assessed using a verbally-administered numerical rating scale (NRS) that ranges from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater pain.
Body pain post-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | Post-biopsy, within 1 minute
  Body pain post-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average body pain during the biopsy procedure, as well as 4) current body pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.
Breast pain post-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | Post-biopsy, within 1 minute
  Breast pain post-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average breast pain during the biopsy procedure, as well as 4) current breast pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.
Body pain 24 hours post-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | 24 hours post-biopsy
  Body pain 24 hours post-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average body pain in the 24 hours post-biopsy, as well as 4) current body pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.
Breast pain 24 hours post-biopsy: Brief Pain Inventory (BPI) Pain Severity Scale | 24 hours post-biopsy
  Breast pain 24 hours post-biopsy will be will be assessed using four questions from the Brief Pain Inventory (BPI) Pain Severity Scale. Women will be asked to rate 1) worst, 2) least, and 3) average breast pain in the 24 hours post-biopsy, as well as 4) current breast pain on a scale from 0 (no pain) to 10 (pain as bad as it could be). Consistent with BPI scoring, items will be averaged to create a composite score that had a possible range of 0 to 10 with higher scores indicating greater pain.

SECONDARY OUTCOMES:
Number of pre-biopsy body pain sites: Body map | Baseline
  To indicate the number of pre-biopsy body pain sites, participants will complete a full body map, indicating the locations of body pain.
Number of pre-biopsy breast pain sites: Breast map | Baseline
  To indicate the number of pre-biopsy breast pain sites, participants will complete a breast map (showing the chest, shoulders, and upper arms), indicating the locations of breast pain.
Anticipated body pain: Anticipatory body pain scale | Baseline
  Prior to biopsy, one question will be asked to assess anticipated body pain (i.e., "How much body pain do you think you will experience during the biopsy today?") on a scale from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater anticipated pain.
Anticipated breast pain: Anticipatory breast pain scale | Baseline
  Prior to biopsy, one question will be asked to assess anticipated breast pain (i.e., "How much breast pain do you think you will experience during the biopsy today?") on a scale from 0 (no pain) to 10 (pain as bad as it could be) with higher scores indicating greater anticipated pain.
Anxiety pre-biopsy: State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) | Baseline
  The State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) will assess the degree of anxiety pre-biopsy. Participants will rate each of the 20 items on a 5-point Likert scale, ranging from 1 (not at all) through 4 (very much). Items will be summed, creating a total score (possible range: 20-80).
Likelihood of cancer pre-biopsy: Likelihood of cancer scale | Baseline
  Likelihood of cancer will be assessed pre-biopsy using a 1 single-item scale. Participants will be asked to indicate what they were told regarding the likelihood of cancer from their recommending radiologist on a scale from 0 (not applicable - they did not discuss this with me) to 5 (high likelihood of cancer) with higher scores indicating a greater likelihood of cancer.
Pain coping strategies pre-biopsy: Coping Strategies Questionnaire (CSQ) | Baseline
  To assess the use of pain coping strategies pre-biopsy, participants will complete the 14-item Coping Strategies Questionnaire (CSQ). Participants will rate how frequently they use seven pain coping strategies (two items per scale) on a scale ranging from 0 (not at all) to 6 (a lot). Items will be averaged, giving a total score on each scale ranging from 0 to 6 with higher scores indicating greater use of pain coping strategies.
Self-efficacy for pain and anxiety pre-biopsy: Self-efficacy for pain and anxiety scale | Baseline
  To assess self-efficacy for managing pain and anxiety pre-biopsy, participants will complete a 4-item scale. Items will be rated on a 10-point scale from 1 (not certain) to 10 (very certain). Items will be averaged to create a composite score, ranging from 0 to 10 with higher scores indicating greater self-efficacy.
Blood pressure pre-biopsy | Baseline
  Blood pressure (systolic/diastolic) pre-biopsy will be measured using an MRI-compatible blood pressure cuff.
Pulse pre-biopsy | Baseline
  Heart rate pre-biopsy will be measured using an MRI-compatible pulse oximeter.
Blood pressure after positioning on the MRI table | After positioning on the MRI table, within 1 minute
  Blood pressure (systolic/diastolic) after positioning on the MRI table will be measured using an MRI-compatible blood pressure cuff.
Pulse after positioning on the MRI table | After positioning on the MRI table, within 1 minute
  Heart rate after positioning on the MRI table will be measured using an MRI-compatible pulse oximeter.
Blood pressure after introducer insertion | After last introducer insertion, within 1 minute
  Blood pressure (systolic/diastolic) after the last introducer is inserted will be measured using an MRI-compatible blood pressure cuff.
Pulse after after introducer insertion | After last introducer insertion, within 1 minute
  Heart rate after the last introducer is inserted will be measured using an MRI-compatible pulse oximeter.
Blood pressure after introducer sheath removal | After last introducer sheath removal, within 1 minute
  Blood pressure (systolic/diastolic) after the last introducer sheath is removed will be measured using an MRI-compatible blood pressure cuff.
Pulse after introducer sheath removal | After last introducer sheath removal, within 1 minute
  Heart rate after the last introducer sheath is removed will be measured using an MRI-compatible pulse oximeter.
Anxiety post-biopsy: State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) | Post-biopsy, within 1 hour
  The State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) will assess the degree of anxiety post-biopsy. Participants will rate each of the 20 items on a 5-point Likert scale, ranging from 1 (not at all) through 4 (very much). Items will be summed, creating a total score (possible range: 20-80).
Likelihood of cancer post-biopsy: Likelihood of cancer scale | Post-biopsy, within 1 hour
  Likelihood of cancer will be assessed post-biopsy using a single-item scale. Participants will be asked to indicate what they were told regarding the likelihood of cancer from the radiologist performing the biopsy on a scale from 0 (not applicable - they did not discuss this with me) to 5 (high likelihood of cancer).
Distraction from pain during biopsy: Attention to pain scale | Post-biopsy, within 1 hour
  Using a 2-item self-report measure, participants will rate 1) the amount of attention they paid to the pain during biopsy and 2) the extent to which they were able to distract themselves from the pain during biopsy on an 11-point scale, ranging from 0 (not at all) to 10 (very much). An ''attention to pain" score (range -10 to +10) will be calculated by subtracting the ability to distract from pain from the amount of attention to pain. The higher the score, the more attention paid to pain.
Distraction from pain during biopsy: Time spent thinking about pain scale | Post-biopsy, within 1 hour
  Participants will also be asked to rate how much time they spent thinking about pain during the biopsy procedure on an 11-point scale, ranging from 0 (none of the time) to 10 (all of the time).
Relaxation during biopsy: Relaxation numerical rating scale (NRS) | Post-biopsy, within 1 hour
  Participants will be asked to indicate how relaxed they were during the biopsy procedure on a scale, ranging from 0 (not relaxed) to 10 (extremely relaxed).
Relaxation during biopsy: Tension Subscale of the Profile of Mood State Short-Form | Post-biopsy, within 1 hour
  Participants will also be provided with a list of six adjectives (i.e., tense, on-edge, uneasy, restless, nervous, and anxious) from the Tension Subscale of the Profile of Mood State Short-Form and be asked to rate each of the adjectives on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely).
Pain coping strategies post-biopsy: Coping Strategies Questionnaire (CSQ) | Post-biopsy, within 1 hour
  To assess the use of pain coping strategies during the biopsy procedure, participants will complete the 14-item Coping Strategies Questionnaire (CSQ). Participants will rate how frequently they used seven pain coping strategies (two items per scale) during the procedure on a scale ranging from 0 (not at all) to 6 (a lot). Items will be averaged, giving a total score on each scale ranging from 0 to 6 with higher scores indicating greater use of pain coping strategies.
Self-efficacy for pain and anxiety during biopsy: Self-efficacy for pain and anxiety scale | Post-biopsy, within 1 hour
  To assess self-efficacy for managing pain and anxiety during the biopsy procedure, participants will complete a 4-item scale. Items will be rated on a 10-point scale from 0 (not certain) to 10 (very certain). Items will be averaged to create a composite score, ranging from 0 to 10 with higher scores indicating greater self-efficacy.
Anxiety 24 hours post-biopsy: State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) | 24 hours post-biopsy
  The State Anxiety Scale of the State-Trait Anxiety Inventory (STAI) will assess the degree of anxiety 24 hours post-biopsy. Participants will rate each of the 20 items on a 5-point Likert scale, ranging from 1 (not at all) through 4 (very much). Items will be summed, creating a total score (possible range: 20-80).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, Ph.D., Principal Investigator — Duke Psychiatry and Behavioral Sciences
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03877146/ICF_000.pdf